CLINICAL TRIAL: NCT04084327
Title: Immunophenotyping of Acute b Cell Lymphoblastic Leukemia
Brief Title: Immunophenotyping of Acute b Cell Lymphoblstic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, ayat ahmed mohamed, principle investigator, South Egypt Cancer Institute
Other Study IDs: acute b All
Record Dates: First submitted 2018-10-16; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-10

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: stastical analysis — 1-Clinical examination data-Complete Blood Count (CBC).Bone Marrow Aspiration (BMA)-Bone Marrow Biopsy (BMB). (if available)-Immunophenotyping results (IPT).Cytogenetic results

SUMMARY:
To study the immunophenotyping pattern of acute B lymphoblastic leukemia in south Egypt Cancer Institute iand its correlation with disease outcome

DETAILED DESCRIPTION:
study the immunophenotyping pattern of acute B lymphoblastic leukemia in south Egypt Cancer Institute from 2009 -2019 and its correlation with disease outcome

ELIGIBILITY:
Inclusion Criteria:

* New cases admitted to SECI Who didn't receive treatment.Age above 1 years old.

Exclusion Criteria:

* Cases who received treatment Patients below 1 years old.Patients diagnosed as AML or T-ALL

Ages: 12 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: new cases Who didn't receive treatment.Age above 1 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival outcome | 10 years
  overall survival outcome
Disease-free survival outcome | 10 years
  Disease-free survival outcome
association of novel CD markers with old markers for assessment of disease outcome | 10 years
  association of novel CD markers with old markers for assessment of disease outcome

REFERENCES:
- [Background] Keegan A, Charest K, Schmidt R, Briggs D, Deangelo DJ, Li B, Morgan EA, Pozdnyakova O. Flow cytometric minimal residual disease assessment of peripheral blood in acute lymphoblastic leukaemia patients has potential for early detection of relapsed extramedullary disease. J Clin Pathol. 2018 Jul;71(7):653-658. doi: 10.1136/jclinpath-2017-204828. Epub 2018 Mar 27. PMID 29588374